CLINICAL TRIAL: NCT01448798
Title: Prospective Randomized Investigation of Athermal Nerve-sparing During Robotic-assisted Laparoscopic Prostatectomy Using a Hemostatic Gelatin-thrombin Matrix
Brief Title: Athermal Nerve-sparing During Robotic-assisted Radical Prostatectomy Using a Hemostatic Matrix.
Acronym: AnPro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Axel Haferkamp, Prof. Dr. med. Axel Haferkamp, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AnPro
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: radical prostatectomy; robotic surgery; erectile dysfunction; continence
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gelatine-thrombin matrix (Experimental): Nerves-paring during robotic-assisted laparoscopic prostatectomy is conducted without mono- or bipolar electrocautery and clipping by using a hemostatic gelatine-thrombin matrix.
  Interventions: Procedure: Application of a hemostatic gelatin-thrombin matrix
- Control (Sham Comparator): Nerve-sparing during robotic-assisted radical prostatectomy is conducted with the use of mono- and bipolar electrocautery and surgical clipping.
  Interventions: Procedure: Use of mono- and bipolar electrocautery and surgical clips

INTERVENTIONS:
Procedure: Application of a hemostatic gelatin-thrombin matrix — Hemostatic gelatin-thrombin matrix is used for hemostasis during nerve-sparing dissection of the prostate.
  Arms: gelatine-thrombin matrix
Procedure: Use of mono- and bipolar electrocautery and surgical clips — Mono- and bipolar electrocautery and surgical clips are used for hemostasis during nerve-sparing dissection of the prostate.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the use of a hemostatic gelatine-thrombin matrix during athermal nerve-sparing prostate resection compared to conventional hemostasis using electrocautery in patients with localized prostate cancer and to investigate effects on postoperative erectile function and continence.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18
* Histologically proven prostate cancer ( Gleason <8; PSA<10ng/ml)
* Disease confined to prostate in clinical examination
* Preoperative IEEF-5-Score>20
* Patient is able to give informed consent

Exclusion Criteria:

* ASA IV-V
* Prior extensive abdominal surgery
* Signs for metastatic disease
* Known allergy against bovine material
* Patient is unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative erectile function | 12 months
  Postoperative erectile function compared to preoperative status assessed validated questionnaires.

SECONDARY OUTCOMES:
Postoperative continence | 12 months
  Postoperative continence compared to preoperative status assessed by validated questionnaires.
Intraoperative bloodloss | During surgery
  Amount of blood collected in the suction during surgery.
Intra- and postoperative complications | Perioperative period
  Intra- and postoperative complications associated to the study´s intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Haferkamp, Prof., Principal Investigator — Johann Wolfgang Goethe University Hospitals, Germany
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt/M., Germany